CLINICAL TRIAL: NCT05628571
Title: Clinical Research Study to Evaluate the Antibacterial Effect 12 Hours After 4-week Use of a Toothpaste Containing Amine Base, Sodium Fluoride and Zinc Lactate
Brief Title: Evaluation of the Antibacterial Effect of a Toothpaste Containing Zinc Lactate
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Colgate Palmolive (Industry); Associação Latinoamericana para Promoção de Saúde Bucal e Pesquisa Odontológica (LAOHA) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CRO-2022-05-MC-MD-BZ-BS
Record Dates: First submitted 2022-11-07; First posted 2022-11-28 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-11

CONDITIONS: Oral Bacterial Infection
Keywords: toothpastes; fluoride; antimicrobial effect; oral bacteria; mucin; zinc
MeSH Terms: conditions — Medullary cystic kidney disease 1 | interventions — green tea bioflavonoid, zinc ascorbate-containing toothpaste

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization lists will be kept confidential by the Investigator, inside a locked cabinet. As patients are included by the Examiner at the first visit (T0), the Investigator will make the allocation. The Examiner and other team members, including the Laboratory Technician, will not know the group to which the patient belongs.
  Toothpastes will be covered with white paper to disguise the identity of the product.
  Participants will also not know which group they belong to and which investigational product they are using. To this end, the products will be distributed in a separate area of the exam room by the Assistant, without the other participants being present.
  The samples will also be labeled with the information of the participant's first and last name initials, the randomization code and the sample collection data (type, intraoral location and collection date). The Laboratory Technician will not know which group the sample belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoride toothpaste (Placebo Comparator): Participants will brush their teeth with a commercially available Fluoride toothpaste (1450 ppm F) and a commercially available adult soft bristle toothbrush
  Interventions: Combination Product: Fluoride Toothpaste
- Zinc toothpaste (Experimental): Participants will brush their teeth with a toothpaste containing amine base, zinc lactate and fluoride (1400 ppm F) and a commercially available adult soft bristle toothbrush
  Interventions: Combination Product: Zinc toothpaste

INTERVENTIONS:
Combination Product: Zinc toothpaste — Participants will brush their teeth with a commercially available, soft-bristle adult toothbrush and toothpaste containing amine-based zinc lactate (0.1%) and fluoride (1400 ppm F).
  Arms: Zinc toothpaste
Combination Product: Fluoride Toothpaste — Participants will brush their teeth with a commercially available, soft-bristle adult toothbrush and toothpaste containing fluoride (1450 ppm F).
  Arms: Fluoride toothpaste

SUMMARY:
The aim of this study is to evaluate the antibacterial effect 12 hours after 4-week use of a toothpaste containing amine base, zinc lactate, and fluoride. For this, healthy people will be invited to use two different toothpaste: control - containing only fluoride; test - containing fluoride plus a combination with zinc. The primary outcome is the efficacy of the test toothpaste in the oral bacterial load reduction in samples of saliva and oral mucosa (obtained through scraping); the second outcome is effect of the test toothpaste in the expression of mucin in the oral mucosa.

DETAILED DESCRIPTION:
Study Design This is a phase III, randomized, single center, parallel-group, double-blind clinical study to evaluate the antibacterial effect of a toothpaste containing an amine, zinc lactate, and fluoride base.

Primary Objective The objective of this study is to evaluate the antibacterial effect 12 hours after using a toothpaste containing amine, zinc lactate and fluoride for 4 weeks.

Secondary Objectives The secondary objective will be to evaluate the impact of a toothpaste containing amine, zinc lactate and fluoride in the quantification of mucin on the surface of the oral mucosa.

Study Intervention Design: Parallel Product Assignment: Randomization Number of individuals: 130 Individuals by age group: 18 to 70 Number of test groups: 2 Treatment regimen: Brushing of the entire mouth with test toothpaste Blind Mode: Double-blind Number of exposures (uses): Twice a day, unattended Study duration: 6 weeks Washout period: Yes Duration of each exposure: 2 minutes of brushing

Study Groups:

1) Test Group: Toothpaste containing amine base, zinc lactate and fluorine (1400 ppm F).

C

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ages 18-70, inclusive;
2. Subjects are available during study duration;
3. Subject is in good general health;
4. A minimum of 15 natural teeth with facial and lingual scorable surfaces, excluding third molars.
5. A willingness to read, understand, and sign the Informed Consent Form after the nature of the study has been fully explained to them.
6. Subjects with baseline whole mouth scores of dental plaque of 1.5 or more and gingivitis index of 1.0 or more.

Exclusion Criteria:

1. Participation in any other clinical study or test panel including clinical studies with oral hygiene formulations within the one month prior to entry into the study.
2. History of dental prophylaxis or treatments in the past month or during study duration.
3. History of medical treatments (e.g: antibiotic, anti-inflammatory, anticoagulant, etc.) during the month preceding study enrollment.
4. Subjects scheduled for any medical procedure during the course of the study.
5. Difficulty complying with study procedures and examinations such as excessive gagging during oral assessment etc.
6. History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses. Allergies to personal care/consumer products or their ingredients.
7. History of diabetes, hepatic, renal disease, inflammatory conditions or transmittable diseases, e.g. heart disease or AIDS.
8. History of rheumatic fever or medical conditions that require prophylactic antibiotics coverage prior to dental procedures.
9. Presence of oral lesions.
10. History of active or severe periodontal disease (PD > 4) and loose teeth.
11. Gross dental caries, severe generalized cervical abrasion and/or enamel abrasion, large fractured or temporary restorations (based on visual examinations).
12. Fixed or removable orthodontic appliances or removable partial dentures.
13. Current smokers and subjects with a history of alcohol or drug abuse.
14. Use of phenolic flavored products, such as mint flavored candies and chewing gum, during the study period.
15. Unable to refrain from oral hygiene for twelve (12) hours prior to scheduled visits.
16. Positive Coronavirus Disease 2019 test 48 hours prior to the screening visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of oral bacteria load | Baseline (previously of the interventions) and after 4 weeks of the interventions
  analysis of oral bacterial load (log10 colony-forming unit/mL) in saliva and oral mucosa biofilm samples, performed by microbial culture

SECONDARY OUTCOMES:
Change of mucin expression in oral mucosa samples | Baseline (previously of the interventions) and after 1, 2, 3 and 4 weeks of the interventions
  quantification of mucin expression produced by the mucin gene (pg/mL) present in samples of the jugal mucosa, performed by means of an ELISA immunoenzymatic test.

IPD SHARING:
Plan to Share IPD: No
All study data will be recorded on forms provided by the sponsor. Only the Investigator, Examiner and Assistant may make entries on the forms. Source data will be retained by the study site. Record security will include keeping written forms in locked and/or sealed file cabinets and/or labeled storage boxes located in a locked room. Access will be denied to all persons except the Principal Investigator and his designees.

REFERENCES:
- [Background] Aguirre A, Mendoza B, Levine MJ, Hatton MN, Douglas WH. In vitro characterization of human salivary lubrication. Arch Oral Biol. 1989;34(8):675-7. doi: 10.1016/0003-9969(89)90024-1. PMID 2597059
- [Background] Ben Lagha A, Yang Y, Trivedi HM, Masters JG, Grenier D. A Dual Zinc plus Arginine formulation attenuates the pathogenic properties of Porphyromonas gingivalis and protects gingival keratinocyte barrier function in an in vitro model. J Oral Microbiol. 2020 Aug 4;12(1):1798044. doi: 10.1080/20002297.2020.1798044. PMID 32944154
- [Background] Carda-Dieguez M, Moazzez R, Mira A. Functional changes in the oral microbiome after use of fluoride and arginine containing dentifrices: a metagenomic and metatranscriptomic study. Microbiome. 2022 Sep 28;10(1):159. doi: 10.1186/s40168-022-01338-4. PMID 36171634
- [Background] Creeth JE, Karwal R, Hara AT, Zero DT. A Randomized in situ Clinical Study of Fluoride Dentifrices on Enamel Remineralization and Resistance to Demineralization: Effects of Zinc. Caries Res. 2018;52(1-2):129-138. doi: 10.1159/000479823. Epub 2018 Jan 5. PMID 29301123
- [Background] Delgado E, Garcia-Godoy F, Montero-Aguilar M, Mateo LR, Ryan M. A Clinical Investigation of a Dual Zinc plus Arginine Dentifrice in Reducing Established Dental Plaque and Gingivitis Over a Six-Month Period of Product Use. J Clin Dent. 2018 Sep;29(Spec No A):A33-40. PMID 30620869
- [Background] Kindblom C, Davies JR, Herzberg MC, Svensater G, Wickstrom C. Salivary proteins promote proteolytic activity in Streptococcus mitis biovar 2 and Streptococcus mutans. Mol Oral Microbiol. 2012 Oct;27(5):362-72. doi: 10.1111/j.2041-1014.2012.00650.x. Epub 2012 May 25. PMID 22958385
- [Background] Manus LM, Daep CA, Begum-Gafur R, Makwana E, Won B, Yang Y, Huang XY, Maloney V, Trivedi HM, Wu D, Masters JG. Enhanced In Vitro Zinc Bioavailability through Rational Design of a Dual Zinc plus Arginine Dentifrice. J Clin Dent. 2018 Sep;29(Spec No A):A10-19. PMID 30620866